CLINICAL TRIAL: NCT05286580
Title: Standardization of Non-academic Center Surgical Morbidity and Mortality Conference: a Type I Hybrid Implementation Non-clinical Trial.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We lost some staffing and were unable to continue the study.
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Lacey LaGrone, Investigator, Poudre Valley Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0261
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Surgery; Surgery--Complications
Keywords: Morbidity and mortality conference; Quality Improvement; Implementation Science
MeSH Terms: interventions — Morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): o Sequential deployment of standardized M&M toolkit at a regional M&M conference.
  Interventions: Behavioral: Morbidity and mortality conference toolkit

INTERVENTIONS:
Behavioral: Morbidity and mortality conference toolkit — * Standardized slide deck
  * Code of conduct
  * Conference planning checklist
  * Case documentation form

SUMMARY:
* Specific Aim 1: Determine impact of standardized morbidity and mortality (M&M) toolkit on provider satisfaction with, and perceived impact of, M&M conference.
* Specific Aim 2: Identify barriers and facilitators to toolkit implementation.

DETAILED DESCRIPTION:
Design:

- Pre-, post- intervention mixed-methods trial.

* Inclusion:

  o M&M conference attendees at enrolled level II and III trauma centers, inclusive of trainees, administrative staff, providers.
* Exclusion:

  * Age < 18
  * Anticipated attendance at <= one M&M conference at study site.
* Intervention:

  * Brief didactic regarding evidence base for M&M conferences.
  * Sequential deployment of standardized M&M toolkit
* Standardized slide deck
* Code of conduct
* Conference planning checklist
* Case documentation form
* Recruitment:

  o Pre/post survey:
* M&M attendees will be invited to scan a QR code made available at the beginning of an M&M conference, and to take 5 minutes to fill the associated survey if they consent.

  o Semi-structured interview:
* The research coordinator contact information will be emailed to M&M listserv, requesting interested parties contact them to schedule an interview.
* Data collection

  o Specific Aim 1:
* Pre/post 10 question digital, anonymous mixed-methods (one free text question) survey

  • Demographics collected: occupation (surgeon / app / non-surgeon physician / other), years in practice (<10, 10-20, >20)
* Observation of M&M to capture:

  • # of attendees
  * # of cases presented at each conference
  * # of cases which include literature review
  * # of cases which include determination of recommended system change (just culture..?)

    * Specific Aim 2:
* Three, six and nine months after initial toolkit deployment we will conduct semi-structured interviews regarding implementation barriers and facilitators.

  * Interviews will be conducted in-person and audio-recorded.
  * Interview guide will be modified to emphasize opportunities for improvement identified in initial quantitative data collection.

    * For instance, if baseline data suggests case referral is the primary problem, will triage discussion of this portion of the M&M process higher and ask additional detail regarding perceived means of improvement.
    * The interview guide scope will not change from that submitted, the emphasis will pivot as described.
  * Data analysis will be ongoing, and results of each interview set will be used to inform adaptation of implementation approach.
* Consent

  o Would like to submit a request for waiver of written consent and inclusion of information sheet in survey with confirmation of understanding but without signature, collection of names.
* Timeline

  o Baseline survey and observational data collection Feb - April 2022, intervention deployment March - May 2022, follow-up data collection Feb - April 2023.
* Study Sites o Northern Colorado M&M (Greeley, Longs Peak, Poudre Valley, Medical Center of the Rockies)

ELIGIBILITY:
Inclusion Criteria:

* M&M conference attendees at enrolled level II and III trauma centers, inclusive of trainees, administrative staff, providers.

Exclusion Criteria:

* Age < 18
* Anticipated attendance at <= one M&M conference at study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Perception of effective M&M conference | one year
  Participant endorses having seen a change at their institution attributable to a discussion at an M&M conference

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No